CLINICAL TRIAL: NCT06640790
Title: Effect of Endodontic Case Difficulty on Endodontic Mishaps: Clinical Study
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Arzu Kaya Mumcu, Assistant professor, Kutahya Health Sciences University
Other Study IDs: KutahyaHSU-1
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Effect of Endodontic Case Difficulty on Endodontic Mishaps; Root Canal Treatment
Keywords: Case Difficulty, Endodontic Mishaps, Postgraduate Dental Education, Root Canal Treatment
MeSH Terms: interventions — Diagnosis-Related Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Case Group — Root canal treated were categorized based on the AAE case difficulty assessment form. Endodontic mishaps investigated included over-instrumentation, working length loss, underfilling, overfilling, apical transportation, instrument fracture, and perforation.

SUMMARY:
The aim of this study investigate the influence of endodontic case difficulty, as categorized by the American Association of Endodontists (AAE) assessment form (low, moderate, high), on the incidence of endodontic mishaps and treatment visit requirements in postgraduate dental students.

ELIGIBILITY:
Inclusion Criteria:

* Primary root canal treatment
* Retreatment

Exclusion Criteria:

* Patients who do not accept to participate to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who refer to our clinic for routine endodontic treatment
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Case difficulty category | Radiographic images were taken at the final treatment appointment. Case difficulty classification of cases was performed according to AEE case difficulty form data, and all radiographs were evaluated in terms of endodontic mishaps within 24 hours.
  The American Association of Endodontists (AAE) has developed a case difficulty form to categorize endodontic cases into three levels: minimal, moderate, and high. This form encompasses three sections: general health status, diagnostic and treatment status, and contributing factors such as trauma, previous treatment, and periodontal disease.
Endodontic mishaps | Radiographic images were taken at the final treatment appointment. Case difficulty classification of cases was performed according to AEE case difficulty form data, and all radiographs were evaluated in terms of endodontic mishaps within 24 hours.
  Endodontic mishaps were classified as follows: over-instrumentation, underfilling (≥2 mm from the radiographic apex), overfilling (≥2 mm from the radiographic apex), canal transportation, instrument separation, lateral or strip perforation.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kaya Mumcu A, Corak M, Kurnaz S, Kiraz G. Effect of endodontic case difficulty on endodontic mishaps and the number of treatment visits: a clinical study. BMC Med Educ. 2025 Dec 9;26(1):63. doi: 10.1186/s12909-025-08437-4. PMID 41366378